CLINICAL TRIAL: NCT04530461
Title: Serologic Profile of SARS CoV2 in COVID-19 Patients With Systemic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: faida agili (Other)
Collaborators: UR17DN02 : Autoimmune Diseases Research Unit (Unknown)
Responsible Party: Sponsor-Investigator, faida agili, Director of Autoimmune Diseases Research Unit (UR17DN02) and Professor in internal medicine departement. Sponsor and Principal Investigator, Military Hospital of Tunis
Organization: Military Hospital of Tunis (Other)
Other Study IDs: UR17DN02-002
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: SARS-CoV Infection; Systemic Disease; Systemic Lupus Erythematosus; Sjogren's Syndrome; Sarcoidosis; Inflammatory Myopathy; Behçet Disease; Rheumatoid Arthritis; Spondyloarthritis
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Sarcoidosis; Myositis; Behcet Syndrome; Arthritis, Rheumatoid; Spondylarthritis | interventions — Serologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serological test — Positive serological test of SARS Cov2

SUMMARY:
An observational study aiming to assess the serological profile of SARS-Cov2 patients with systemic diseases such as systemic lupus erythematosus, Sjogren syndrome, sarcoidosis, inflammatory myopathies, Behçet's disease, Rheumatoid arthritis and Spondyloarthritis

DETAILED DESCRIPTION:
The study is a prospective, observational, multicenter clinical trial to be conducted in the internal medicine, rheumatology and virology departments of Military Hospital of Tunis. After obtaining informed consent from the patient, the investigator will perform an inclusion visit made of a patient interview and performing blood sample to search for IgG and anti-SARS IgM CoV2.

Patients with IgM-like antibodies will have an RT-PCR test for active infection. If the study participants will be diagnosed with COVID-19 positive during the study period, the attending physician is entitled to decide on their management based on the severity of the clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* One of the following conditions: systemic lupus, Sjögren's syndrome, rheumatoid arthritis, inflammatory myopathies, spondyloarthritis, sarcoidosis and Behçet's disease.
* Informed consent obtained and signed

Exclusion Criteria:

* Refusal to repeat blood sampling if the first one was badly performed
* Informed consent not obained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with one of the following conditions: systemic lupus, Sjögren's syndrome, rheumatoid arthritis, inflammatory myopathies, spondyloarthritis, sarcoidosis and Behçet's disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Serological Profile | Inclusion
  Number of patients with positive serological test of SARS Cov2

CONTACTS AND LOCATIONS:
Overall Officials: Faida Ajili, MD, Study Chair — Military Hospital of Tunis
Locations (1):
- Military Hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No